CLINICAL TRIAL: NCT05704413
Title: Digestive Biobank for Exploring Microbiota-host Interactions
Acronym: BiomHost
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180540
Record Dates: First submitted 2019-02-18; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Colorectal Cancer; Indeterminate Colitis
Keywords: Microbiota; inflammatory bowel disease; Crohn's disease; ulcerative colitis; colorectal cancer; post-operative cognitive disorders; mood disorders; immune system.
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Colorectal Neoplasms; Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Intestinal surgical waste: Surgical samples will be rinsed in saline and aliquoted in dry tubes (minimum 5 aliquots) and lateral RNA (minimum 3 aliquots) and then frozen at -80°C
  * Intestinal contents: They will be aliquoted (at least 5 aliquots) in dry tubes for freezing at -80°C
  * blood samples (1 dry tube and 2 EDTA tubes of 7ml): centrifigation and aliquoting of serum and plasma, storage at -80°C
  * whole blood samples (1 sodium heparin tube of 5ml) : stimulation and fixation with proteomic stabilizer, storage at -80°
  * DNA ; Stored at -20°C
  * stools: aliquoting and storage at -80°C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- digestive cancer or IBD: Patient with digestive cancer or IBD having surgery with intestinal resection planned in the Visceral Surgery Department of St Antoine Hospital

SUMMARY:
Constitution of a biobank of tissues, whole blood and plasma samples and stools to identify markers associated with treatment response, postoperative morbidity including neuro-cognitive and mood complications and prognosis of Inflammatory Bowel disease or colorectal cancer.

DETAILED DESCRIPTION:
Inflammatory Bowel disease (Crohn, Ulcerative colitis) and colorectal cancer are frequent affections and the microbiota plays a major role in their physiopathology involving the immune system. In this setting, the interplay between gut microbiota and brain is still unexplored.

To evaluate the interaction of the microbiota and the immune system with the host in these two chronic diseases, we aim to create a prospective biobank.

A small amount of tissue will be taken during surgery. A whole blood, plasma and stoll samples will also be taken from the patient.

All samples will be anonymized.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis, Crohn's disease or colorectal disease
* Digestive resection with useless tissue available
* Information consent signed

Exclusion Criteria:

- Patients < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years-old. With an Ulcerative colitis, Crohn's Disease or colorectal cancer Operated in the Departement of digestive surgery of Saint-Antoine Hospital After signature of the information consent
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Relation between biological parameters and outcomes of digestive disease (IBD, CRC) | up to 12 months after the incusion
  identify relations between serumon response to treatment, postoperative outcomes including neuro-cognitive and mood complications and prognosis.

SECONDARY OUTCOMES:
Relation between biological parameters and outcomes of digestive disease (IBD, CRC) | up to 12 months after the incusion
  identify relations between plasma on response to treatment, postoperative outcomes including neuro-cognitive and mood complications and prognosis.
Relation between biological parameters and outcomes of digestive disease (IBD, CRC) | up to 12 months after the incusion
  identify relations between DNA on response to treatment, postoperative outcomes including neuro-cognitive and mood complications and prognosis.
Relation between biological parameters and outcomes of digestive disease (IBD, CRC) | up to 12 months after the incusion
  identify relations between faeces) on response to treatment, postoperative outcomes including neuro-cognitive and mood complications and prognosis.
Exploratory study on the physiopathology of host-microbiota interactions to determinate the occurrence of intestinal and extra-intestinal complications | up to two months after the incusion
  genetic polymorphisms, serum markers, intestinal microbiota markers to determining the occurrence of intestinal and extra-intestinal complications
Exploratory study on the physiopathology of host-microbiota interactions to determinate the response to treatments | up to two months after the incusion
  genetic polymorphisms, serum markers, intestinal microbiota markers determining : response to treatments
Exploratory study on the physiopathology of host-microbiota interactions | up to two months after the incusion
  genetic polymorphisms, serum markers, intestinal microbiota markers determining : interactions between host and microbiota
Brain-microbiota interaction | up to two months after the incusion
  Exploring the pathophysiology of host-microbiota interactions in postoperative cognitive or behavioral changes involving inflammation pathways

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie LEFEVRE, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Chirurgie Viscérale - Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided